CLINICAL TRIAL: NCT02846753
Title: Implantation of the Venus P-Valve™ in the Pulmonic Position in Patients With Native Outflow Tracts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Venus MedTech (HangZhou) Inc. (Industry)
Collaborators: IQVIA Inc. (Industry); TheraGenesis (Unknown); Intrials (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMT-001CE
Record Dates: First submitted 2016-05-03; First posted 2016-07-27 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Regurgitation
MeSH Terms: conditions — Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation of Venus P-Valve™ (Experimental): Implantation of the Venus P-Valve™ in the pulmonic position in patients with native outflow tracts; trans catheter heart valve replacement.
  Interventions: Procedure: trans catheter heart valve replacement

INTERVENTIONS:
Procedure: trans catheter heart valve replacement — trans catheter heart valve replacement

SUMMARY:
A prospective, non-randomized multi-center clinical investigation of the Venus P-Valve™ for the treatment of pulmonary regurgitation with or without stenosis in patient with native outflow tracts.

DETAILED DESCRIPTION:
This study evaluates the implantation of the Venus P-Valve™ for the treatment of patients with an incompetent pulmonic valve, which causes blood to flow back from the pulmonary artery into the right heart ventricle during pumping of the heart (pulmonary regurgitation). Patients with and without narrowing (stenosis) of the right ventricular outflow tract will be included. The purpose of this protocol is to assess the safety and performance of Venus P-Valve™ implantation.

Post-procedure, a clinical visit will be scheduled at 30 days, 6 month, 12 months, and annually thereafter to 3 years. Population: Patients≥12 years with a body weight of ≥30kg, with significant pulmonary regurgitation (≥3+) with or without right ventricular outflow tract (RVOT) stenosis (mean Doppler gradient ≥35mmHg) with native right ventricular outflow tracts.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet all of the following Inclusion criteria:

* Age: range from 12-70 years of age
* Weight must be "equal to" or exceed 30 kilograms
* Subject presents with evidence of moderate or severe (≥3+) pulmonary regurgitation by TTE
* Subject presents with >30% pulmonary regurgitation fraction as defined by cardiac MRI
* Subject is symptomatic from his/her pulmonary regurgitation or meets MRI criteria for intervention: right ventricular ejection fraction (RVEF) < 45%, pulmonary regurgitant fraction (PRRF) >30% and increased right ventricular end-diastolic volume (RVEDV) >150ml/m2
* Subject will comply with specified follow-up evaluations, including echocardiograms and MRI
* The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the ethics committee and regulatory authority if applicable of the respective clinical site
* The subject and the treating physician agree that the subject will return for all required post-procedure follow up visits
* Catheterization is determined to be feasible by the treating physician

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

* Active infection requiring current antibiotic therapy (if temporary illness, subject may be a candidate 4 weeks after discontinuation of antibiotics)
* Severe chest wall deformity
* Leukopenia (WBC<3000 mm3)
* Acute or chronic anemia (Hb <90g/l)
* Platelet count <100,000 cells/mm3
* In the judgment of the investigator, percutaneous introduction and delivery of the valve is not feasible
* Need for emergency cardiac or vascular surgery, including pulmonary embolectomy, for any reason
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
* History of, or active, endocarditis, unless the endocarditis has been treated >6 months previous to the procedure
* History of or current intravenous drug abuse
* A known hypersensitivity to aspirin or heparin
* Currently participating in an investigational drug or another device study [Note: Trials requiring extended follow up for products that were investigational, but have since become commercially available, are not considered investigational devices.]
* Major or progressive non-cardiac disease resulting in a life expectancy of <1yr
* Obstruction of the central veins preventing advancement of the pulmonary bioprosthesis delivery system to the heart
* Positive urine or serum pregnancy test in female subjects of child-bearing potential
* Ileofemoral vessel characteristics that would preclude safe placement of 19 French (F), 22 F and 24 F introducer sheath
* Contraindication for cardiac magnetic resonance imaging or inability to cooperate with a cardiac magnetic resonance imaging exam
* Need for concomitant interventional procedures

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Venus P-Valve™ measured as probability of death/reoperation | month 12 follow-up
  Occurrence of death or reoperation (Valve and/or procedure related) calculated as a composite freedom-of-death and -reoperation probability at 12 months. The acceptance criterion for mortality and reoperation is 16% (or equivalently 84% freedom from death and reoperation). If the lower 95% confidence limit for survival and freedom from reoperation at 12 months is greater than 84%, the acceptance criterion for safety will have been met.
Safety of Venus P-Valve™ measured as probability of Major Adverse Cardiac and Cerebro-vascular Event (MACCE) | month 1 follow-up
  Occurrence of MACCE (defined as death, myocardial infarction, reoperation, vascular injury resulting in the need for an unplanned vascular grafting intervention, stroke, and pulmonary embolism) calculated as freedom-from-MACCE probability at month-1, calculated using the Kaplan Meier method
Performance of Venus P-Valve™ measured as Success rate of valve placement and implantation | up to 30 days
  The device success is defined as the percentage of subjects with successful implant of the P-Valve assessed at the earliest evaluable echocardiogram. Linearized rates will be presented.
Hemodynamic Performance of Venus P-Valve™ measured as the mean transvalvular pressure (mmHg) | 1 month
  Hemodynamic performance, measured as the mean transvalvular pressure gradient measured by transthoracic echocardiogram at month-1
Performance of Venus P-Valve™ measured as change of pulmonary regurgitation (regurgitation classification by MRI) | baseline and month 6
  Improvement or abolition of pulmonary regurgitation assessed by MRI at baseline and month 6, with grading of pulmonary stenosis defined as: mild <2, moderate: 2-4; severe >4
Performance of Venus P-Valve™ measured as change of pulmonary regurgitation (regurgitation classification by transthoracic echocardiogram) | baseline, day 1, month 1, 6, 12 and annually thereafter to 3 years post procedure
  Improvement or abolition of pulmonary regurgitation assessed by transthoracic echocardiogram at baseline, day 1, month 1, 6, 12 and annually thereafter to 3 years post procedure, with grading of pulmonary stenosis defined as: mild <2, moderate: 2-4; severe >4
Performance of Venus P-Valve™ measured as percentage of subjects with structural valve deterioration | month 6
  Structural valve deterioration assessment includes stent fracture, leaflet mobility, thickening and calcification

SECONDARY OUTCOMES:
Safety measured as percentage of subjects experiencing serious adverse events | up to third year of follow-up
  Within the duration of the study of the percentage of patients experiencing the following events is measured:
  * Device migration/embolization
  * Valvar thrombosis
  * Thromboembolism
  * Bleeding
  * Paravalvar leak
  * Endocarditis
  * Nonstructural dysfunction
  * Explant
  * Hemolysis
  * Arrhythmias
  * all other serious adverse events as defined in protocol section 6.2
Functional improvement measured as decreased pulmonary regurgitation (regurgitation classification by transthoracic echocardiogram ) | 1 month
  Improved valve function demonstrated by a decrease in pulmonary regurgitation (PR) to mild or less (≤ 2) by transthoracic echocardiogram (TTE) at month-1
Functional improvement measured as decreased pulmonary regurgitation (regurgitation classification by MRI) | month 6
  Improved valve function demonstrated by a decrease in pulmonary regurgitation (PR) to mild or less (≤ 2) by MRI at month-6

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel A. Qureshi, MD, Principal Investigator — Evelina Children's Hospital

IPD SHARING:
Plan to Share IPD: No
The results of the study will be reported and disseminated in peer-reviewed scientific journals, internal reports, conference presentations and submissions to regulatory authorities. Nevertheless, all data used in the analysis and reporting of this clinical investigation will be without identifiable reference to individual patients. All the data will be anonymous.